CLINICAL TRIAL: NCT00780884
Title: Influence of Acupuncture on Emotional Measures and Quality of Sleep Among Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0015-08
Record Dates: First submitted 2008-10-26; First posted 2008-10-28 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia; Schizoaffective
Keywords: acupuncture; schizophrenia; insomnia
MeSH Terms: conditions — Schizophrenia; Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- acupuncture needles (Experimental): Acupuncture needles named acuzone needles. The acuzone needles are sterile and single use, manufactured by DONG BANG MEDICAL CO.,LTD.
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — 16 sessions of acupuncture treatment, twice a week.

SUMMARY:
Insomnia, a common feature of schizophrenia, has serious consequences for daytime functioning and quality of life. Although insomnia is most often treated with medication, a growing number of studies have demonstrated the efficiency of a variety of relaxation techniques, cognitive behavioral therapies and alternative medicine procedures. Acupuncture is among the oldest healing practices in the world. Part of traditional Chinese medicine, acupuncture aims to restore and maintain health through the stimulation of specific points on the body. Previous studies have demonstrated that acupuncture has a positive influence on a number of diseases and disorders, among them Depression, Chronic Pain and Sleep Disorders. Hence, the aim of the present study is to examine the effects of acupuncture as a treatment for insomnia in schizophrenic patients.The study begins with a 7-day, running-in, no-treatment period, followes by an 8-week experimental period. During the experimental period, subjects receive acupuncture treatments twice a week. During the first week of the study (no-treatment period) and the last week of the experimental period, subjects' sleep is monitored with a wrist actigraph, and subjects complete a wide spectrum of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. schizophrenia or schizoaffective disorder - diagnosed according DSM-4.
2. capability to sign inform consent.

Exclusion Criteria:

1. unstable physical illness
2. drug or alchohol abuse or dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
sleep efficiency | 8 weeks

SECONDARY OUTCOMES:
anxiety and depression levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Kremer, MD, Principal Investigator — Haemek Mediacl Center
Locations (1):
- Haemek Medical Center, Afula, Israel